CLINICAL TRIAL: NCT05461898
Title: RehabGBs: Rehabilitation in People With Guillain-Barré Syndrome
Acronym: RehabGBs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centro de Reabilitacao do Norte (Other)
Collaborators: Aveiro University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RehabGBs
Record Dates: First submitted 2022-07-06; First posted 2022-07-18 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2024-12

CONDITIONS: Guillain-Barré Syndrome
Keywords: Rehabilitation; Inspiratory Muscle Training
MeSH Terms: conditions — Guillain-Barre Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Inpatient Rehabilitation + Inspiratory Muscle Training (Experimental): * The inpatient rehabilitation program included individualized, functional goal-oriented treatment, with approximately 5 hours of intervention a day, 5 days/week for a total of 6 weeks, with integrated rehabilitation care.
  * The inspiratory muscle training included a 6 weeks intervention with electronic-controlled valve device
  Interventions: Other: Inpatient Rehabilitation; Other: Inspiratory muscle training
- Inpatient Rehabilitation (Active Comparator): - The inpatient rehabilitation program included individualized, functional goal-oriented treatment, with approximately 5 hours of intervention a day, 5 days/week for a total of 6 weeks, with integrated rehabilitation care.
  Interventions: Other: Inpatient Rehabilitation

INTERVENTIONS:
Other: Inpatient Rehabilitation — Standard inpatient rehabilitation program with a interdisciplinary team that included a physiotherapist who ensured muscle strength, balance, aerobic and functional training, an occupational therapist who provided training of basic and instrumental activities of daily living and education of energy conservation techniques and a a speech and language therapist for swallowing training.
Other: Inspiratory muscle training — Inspiratory muscle training protocol during 6 weeks with a electronic-controlled valve device
  Arms: Inpatient Rehabilitation + Inspiratory Muscle Training

SUMMARY:
Guillain-Barré syndrome (GBS) is a neurological disease characterized by an inflammation of peripheral nerves, which might be responsible for long-term disability.

Respiratory muscle weakness is a complication of GBS and might be responsible for respiratory symptoms, inadequate secretion clearance or hypoventilation, with negative impact on daily life.

Inspiratory muscle training has been applied in respiratory and neurological diseases and benefits have been observed in symptoms (e.g., dyspnoea), pulmonary function, exercise capacity and quality of life. Nevertheless, results of this intervention in people with GBS are yet unknown. Moreover, rehabilitation is a key player in the recovery of these highly complex patients, however, the interpretation of the magnitude of its effects has been limited by the absence of minimal clinically important differences for most outcome measures. To overcome these drawbacks, methodologically robust trials are needed to build evidence-based rehabilitation to improve clinical care on GBS.

The primary aim of this project (RehabGBs) is to develop an inspiratory muscle training protocol - InspireGBs and assess its effects on respiratory muscle strength, peak cough flow, pulmonary function, dyspnoea, fatigue, functional status and quality of life in people with GBS, through a randomised controlled trial. Secondary aims are to: i) establish minimal clinically important differences of Functional Assessment of Chronic Illness Therapy-Fatigue Subscale, Medical Research Council - Manual Muscle Testing, Vital capacity, Maximal Inspiratory Pressure, Peak Cough Flow, Functional Independence Measure and Quality of Life for inpatient rehabilitation programmes of people with GBS ii) Evaluate the prevalence of nocturnal hypoventilation in GBS.

DETAILED DESCRIPTION:
Guillain-Barré syndrome (GBS) is an acute inflammatory demyelinating polyradiculoneuropathy and is the most common cause of acute flaccid paralysis. Its annual global incidence is between 0.8 - 1.9 cases per 100,000 people.

GBS is usually preceded by infection or other immune stimulation that induces an aberrant autoimmune response targeting peripheral nerves and their spinal roots. It is characterized by rapid progressive bilateral muscle weakness of the lower limbs and/or arms, in combination with hyporeflexia or areflexia, and most patients reach their maximum disability within 2-4 weeks.Various phenotypes have been described, including acute inflammatory demyelinating polyradiculoneuropathy, acute motor axonal neuropathy, acute motor sensory axonal neuropathy and Miller-Fisher syndrome.

Overall, the clinical course, severity and outcomes of people with GBS are highly heterogeneous. Significant disability, including incomplete recovery of motor (i.e., ambulation) and sensory function, as well as fatigue, pain, respiratory insufficiency and psychological distress might exist after the acute phase. But long-term significant impacts, two years after the onset, on daily activities, work, social activities and health-related quality of life have also been reported. The most often feature is an impairment of the motor capacity, but respiratory muscle weakness is a common complication in people with GBS and may result in decrease vital capacity, chest wall expansion and coughing strength, causing atelectasis and pulmonary infections. Therefore, it is generally accepted that respiratory muscle weakness causes increased morbidity and mortality, owing to the combination of poor airway protection, inadequate secretion clearance and hypoventilation. Previous studies already identified these clinical manifestations in acute GBS. However, prevalence of hypoventilation and inspiratory muscle weakness in subacute phase of GBS is still unknown. Early recognition and treatment of respiratory muscle weakness is important in people with GBS and physiotherapy interventions may be useful to successfully manage these patients.

Inspiratory muscle training (IMT) is a cheap and free of side-effects therapeutic modality, which consists of breathing exercises using a pressure threshold device, that has been applied in several diseases. In patients with chronic obstructive pulmonary disease, IMT improve inspiratory muscle function, exertional dyspnoea and exercise capacity. In patients with neuromuscular disease, has been suggested that IMT increases inspiratory muscle strength and lung volumes, especially in those with muscular dystrophies. In addition, a randomized control trial concluded that IMT in acute patients increases inspiratory muscle strength and quality of life. However, there are no studies about rehabilitation approaches, such IMT, to improve symptoms (i.e. dyspnoea or fatigue), pulmonary function, functional status and quality of life in people with GBS.

Rehabilitation, namely inpatient rehabilitation programmes, is therefore key for the recovery of symptoms, functional outcomes, community participation and quality of life of these highly complex patients. Nevertheless, insufficient high-quality literature, still precludes definitive conclusions about the effects of rehabilitation in people with GBS. Additionally, the interpretation of the magnitude of its effects is challenging due to the lack of minimal clinically important differences (MCIDs) for most outcome measures used in rehabilitation of people with GBS. A MCIDs is the smallest change in a measure that will be perceived as an important improvement for the patient. Such values constitute thresholds for clinical meaningfulness. Therefore, establishing MCIDs is essential to determine effectiveness of rehabilitation and guide clinical decision-making in the management of people with GBS.

In conclusion, by developing and implementing RehabGBs, we will contribute to build evidence-based rehabilitation practices and optimise care in GBS, by: i) assessing the effects of IMT in people with GBS; ii) establishing minimal clinical important differences of rehabilitation outcome measures, to help clinicians better understand the magnitude of the effects of the intervention and determine effectiveness of rehabilitation in people with GBS; iii) evaluate the prevalence of nocturnal hypoventilation in people with GBS.

Therefore, the primary aim of RehabGBs is to:

1. Evaluate, through a randomised controlled trial, the effects of InspireGBs - inspiratory muscle training protocol on respiratory muscle strength, peak cough flow, lung function, dyspnoea, fatigue, functional status and quality of life in people with GBS.

The secondary aims of the project are to:

1. Establish the MCIDs for rehabilitation programmes in people with GBS for Functional Assessment of Chronic Illness Therapy-Fatigue Subscale, Modified Borg Scale, Medical Research Council - Manual Muscle Testing, Vital capacity, Maximal Inspiratory pressure, Peak Cough Flow, Functional Independence Measure and EuroQol Five-Dimensional Questionnaire.
2. Evaluate the prevalence of nocturnal hypoventilation in people with sub-acute GBS.

Study Design & Intervention

InspireGBs is an inspiratory muscle training programme which will be implemented to people with GBS for 6 weeks during an inpatient rehabilitation programme. They will receive IMT for 5 days/week using the PowerBreath KH2. This handheld device applies a constant resistance provided by a electronic-controlled valve. Training will be set initially at a load of approximately 50% of patients' maximal inspiratory mouth pressure. This initial load will be daily increased during the programme based on symptom scores (modified Borg dyspnoea Scale ratings of 4-6 of 10).Total daily training time will consist of 6 cycles of 30 breaths (3 cycles, twice daily).

Patients will be recruited as described and randomly allocated by a computer-generated adaptive random allocation schedule (in a ratio 1:1) to either the experimental or control groups. All participants will receive the inpatient rehabilitation programme. This programme will be tailored to each patient, with approximately 5 hours of intervention/day for 5 days/week (typically for 14 weeks). An interdisciplinary team composed of physiotherapy; occupational therapy; speech and language therapy; and medical, pharmacological, nursery, psychology, clinical dietitian and social worker will be involved, as needed.

Sample Size Estimation

Based on an inspiratory muscle training study conducted in people with spinal cord injury, it is anticipated that a minimum of 64 participants (32 in each group) will be needed to detect a between-group difference of 10 cmH2O in the primary outcome measure (power=80%, α=0.05, 2-tailed). Since in GBS rehabilitation interventions dropout rates are around 15%, 74 participants will be needed.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years
* diagnosed with Guillain Barré Syndrome
* willing to participate in an inpatient rehabilitation program
* able to provide informed consent

Exclusion Criteria:

* presence of significant cardiac and musculoskeletal diseases
* tracheostomized patients
* signs of cognitive impairment or current neoplastic or immunological disease which may preclude their participation in the rehabilitation program and participation in any other therapeutic intervention in addition to standard of care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in maximal inspiratory pressure | 6 weeks
  Respiratory muscle strength will be assessed with maximal respiratory pressure tests

SECONDARY OUTCOMES:
Change in maximal expiratory pressure | 6 weeks
  Respiratory muscle strength will be assessed with maximal respiratory pressure tests
Change in Peak cough flow | 6 weeks
  Peak cough flow is the peak expiratory flow during a cough maneuver and will be measured three times and the best value will be used for analysis, using a hand-held peak flow meter.
Change in Nocturnal transcutaneous carbon dioxide and peripheral oxygen saturation | 6 weeks
  Nocturnal transcutaneous carbon dioxide will be recorded simultaneously for one night using a digital transcutaneous (SenTec, Switzerland)
Change in Medical Research Council - Manual Muscle Testing | 6 weeks
  This test is performed by applying manual resistance and the score is a sum of the strength of six muscle groups: 1) deltoid; 2) biceps; 3) wrist extensor; 4) iliopsoas; 5) quadriceps femoris; and 6) anterior tibial tested bilaterally, from grade 5 (i.e. the patient an move through the full range of motion against gravity and hold an isometric contraction against maximal resistance for 3 seconds) to grade 0 (i.e. no visible contraction)
Change in Functional Assessment of Chronic Illness Therapy-Fatigue Subscale | 6 weeks
  Functional Assessment of Chronic Illness Therapy-Fatigue Subscale is a multidimensional 13-item questionnaire assessing tiredness, weakness, and difficulty in handling daily activities due to fatigue, over the previous 7 days. Scores range from 0 to 52, with higher scores indicating less fatigue.
Change in Functional Independence Measure | 6 weeks
  Functional status will be measured with the Functional Independence Measure, an 18-item clinician reported scale which measures independent performance in self-care, sphincter control, transfers, locomotion, communication, and social cognition. Scores range from 1 to 7 (i.e. 1 = total assistance and 7 = complete independence). The score reflects burden of care in each area measured.

CONTACTS AND LOCATIONS:
Overall Officials: Alda S Marques, PhD, Study Director — School of Health Sciences, University of Aveiro (ESSUA)
Locations (1):
- Centro de Reabilitação do Norte, Vila Nova de Gaia, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leonhard SE, Mandarakas MR, Gondim FAA, Bateman K, Ferreira MLB, Cornblath DR, van Doorn PA, Dourado ME, Hughes RAC, Islam B, Kusunoki S, Pardo CA, Reisin R, Sejvar JJ, Shahrizaila N, Soares C, Umapathi T, Wang Y, Yiu EM, Willison HJ, Jacobs BC. Diagnosis and management of Guillain-Barre syndrome in ten steps. Nat Rev Neurol. 2019 Nov;15(11):671-683. doi: 10.1038/s41582-019-0250-9. Epub 2019 Sep 20. PMID 31541214
- [Background] Willison HJ, Jacobs BC, van Doorn PA. Guillain-Barre syndrome. Lancet. 2016 Aug 13;388(10045):717-27. doi: 10.1016/S0140-6736(16)00339-1. Epub 2016 Mar 2. PMID 26948435
- [Background] van den Berg B, Walgaard C, Drenthen J, Fokke C, Jacobs BC, van Doorn PA. Guillain-Barre syndrome: pathogenesis, diagnosis, treatment and prognosis. Nat Rev Neurol. 2014 Aug;10(8):469-82. doi: 10.1038/nrneurol.2014.121. Epub 2014 Jul 15. PMID 25023340
- [Background] Forsberg A, Press R, Einarsson U, de Pedro-Cuesta J, Holmqvist LW. Disability and health-related quality of life in Guillain-Barre syndrome during the first two years after onset: a prospective study. Clin Rehabil. 2005 Dec;19(8):900-9. doi: 10.1191/0269215505cr918oa. PMID 16323390
- [Background] Green C, Baker T, Subramaniam A. Predictors of respiratory failure in patients with Guillain-Barre syndrome: a systematic review and meta-analysis. Med J Aust. 2018 Mar 5;208(4):181-188. doi: 10.5694/mja17.00552. PMID 29490222
- [Background] van den Berg B, Storm EF, Garssen MJP, Blomkwist-Markens PH, Jacobs BC. Clinical outcome of Guillain-Barre syndrome after prolonged mechanical ventilation. J Neurol Neurosurg Psychiatry. 2018 Sep;89(9):949-954. doi: 10.1136/jnnp-2018-317968. Epub 2018 Apr 7. PMID 29627773
- [Background] Walterspacher S, Kirchberger A, Lambeck J, Walker DJ, Schworer A, Niesen WD, Windisch W, Hamzei F, Kabitz HJ. Respiratory Muscle Assessment in Acute Guillain-Barre Syndrome. Lung. 2016 Oct;194(5):821-8. doi: 10.1007/s00408-016-9929-5. Epub 2016 Aug 9. PMID 27506902
- [Background] Orlikowski D, Prigent H, Sharshar T, Lofaso F, Raphael JC. Respiratory dysfunction in Guillain-Barre Syndrome. Neurocrit Care. 2004;1(4):415-22. doi: 10.1385/NCC:1:4:415. PMID 16174943
- [Background] Aslan GK, Gurses HN, Issever H, Kiyan E. Effects of respiratory muscle training on pulmonary functions in patients with slowly progressive neuromuscular disease: a randomized controlled trial. Clin Rehabil. 2014 Jun;28(6):573-81. doi: 10.1177/0269215513512215. Epub 2013 Nov 25. PMID 24275453
- [Background] Charususin N, Gosselink R, Decramer M, Demeyer H, McConnell A, Saey D, Maltais F, Derom E, Vermeersch S, Heijdra YF, van Helvoort H, Garms L, Schneeberger T, Kenn K, Gloeckl R, Langer D. Randomised controlled trial of adjunctive inspiratory muscle training for patients with COPD. Thorax. 2018 Oct;73(10):942-950. doi: 10.1136/thoraxjnl-2017-211417. Epub 2018 Jun 18. PMID 29914940
- [Background] Boswell-Ruys CL, Lewis CRH, Wijeysuriya NS, McBain RA, Lee BB, McKenzie DK, Gandevia SC, Butler JE. Impact of respiratory muscle training on respiratory muscle strength, respiratory function and quality of life in individuals with tetraplegia: a randomised clinical trial. Thorax. 2020 Mar;75(3):279-288. doi: 10.1136/thoraxjnl-2019-213917. Epub 2020 Jan 14. PMID 31937553
- [Background] Koessler W, Wanke T, Winkler G, Nader A, Toifl K, Kurz H, Zwick H. 2 Years' experience with inspiratory muscle training in patients with neuromuscular disorders. Chest. 2001 Sep;120(3):765-9. doi: 10.1378/chest.120.3.765. PMID 11555507
- [Background] Bissett BM, Leditschke IA, Neeman T, Boots R, Paratz J. Inspiratory muscle training to enhance recovery from mechanical ventilation: a randomised trial. Thorax. 2016 Sep;71(9):812-9. doi: 10.1136/thoraxjnl-2016-208279. Epub 2016 Jun 2. PMID 27257003
- [Background] Simatos Arsenault N, Vincent PO, Yu BH, Bastien R, Sweeney A. Influence of Exercise on Patients with Guillain-Barre Syndrome: A Systematic Review. Physiother Can. 2016;68(4):367-376. doi: 10.3138/ptc.2015-58. PMID 27904236
- [Background] Khan F, Amatya B. Rehabilitation interventions in patients with acute demyelinating inflammatory polyneuropathy: a systematic review. Eur J Phys Rehabil Med. 2012 Sep;48(3):507-22. Epub 2012 Jul 23. PMID 22820829
- [Background] Sulli S, Scala L, Berardi A, Conte A, Baione V, Belvisi D, Leodori G, Galeoto G. The efficacy of rehabilitation in people with Guillain-Barre syndrome: a systematic review of randomized controlled trials. Expert Rev Neurother. 2021 Apr;21(4):455-461. doi: 10.1080/14737175.2021.1890034. Epub 2021 Feb 23. PMID 33567916
- [Background] Malec JF, Ketchum JM. A Standard Method for Determining the Minimal Clinically Important Difference for Rehabilitation Measures. Arch Phys Med Rehabil. 2020 Jun;101(6):1090-1094. doi: 10.1016/j.apmr.2019.12.008. Epub 2020 Jan 15. PMID 31953077
- [Background] Khan F, Pallant JF, Amatya B, Ng L, Gorelik A, Brand C. Outcomes of high- and low-intensity rehabilitation programme for persons in chronic phase after Guillain-Barre syndrome: a randomized controlled trial. J Rehabil Med. 2011 Jun;43(7):638-46. doi: 10.2340/16501977-0826. PMID 21667009
- [Background] Ogna A, Quera Salva MA, Prigent H, Mroue G, Vaugier I, Annane D, Lofaso F, Orlikowski D. Nocturnal hypoventilation in neuromuscular disease: prevalence according to different definitions issued from the literature. Sleep Breath. 2016 May;20(2):575-81. doi: 10.1007/s11325-015-1247-2. Epub 2015 Sep 4. PMID 26338464
- [Background] Bowen DJ, Kreuter M, Spring B, Cofta-Woerpel L, Linnan L, Weiner D, Bakken S, Kaplan CP, Squiers L, Fabrizio C, Fernandez M. How we design feasibility studies. Am J Prev Med. 2009 May;36(5):452-7. doi: 10.1016/j.amepre.2009.02.002. PMID 19362699
- [Background] Laveneziana P, Albuquerque A, Aliverti A, Babb T, Barreiro E, Dres M, Dube BP, Fauroux B, Gea J, Guenette JA, Hudson AL, Kabitz HJ, Laghi F, Langer D, Luo YM, Neder JA, O'Donnell D, Polkey MI, Rabinovich RA, Rossi A, Series F, Similowski T, Spengler CM, Vogiatzis I, Verges S. ERS statement on respiratory muscle testing at rest and during exercise. Eur Respir J. 2019 Jun 13;53(6):1801214. doi: 10.1183/13993003.01214-2018. Print 2019 Jun. PMID 30956204
- [Background] Bach JR, Goncalves MR, Paez S, Winck JC, Leitao S, Abreu P. Expiratory flow maneuvers in patients with neuromuscular diseases. Am J Phys Med Rehabil. 2006 Feb;85(2):105-11. doi: 10.1097/01.phm.0000197307.32537.40. PMID 16428900
- [Background] Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. Standardisation of spirometry. Eur Respir J. 2005 Aug;26(2):319-38. doi: 10.1183/09031936.05.00034805. No abstract available. PMID 16055882
- [Background] Kleyweg RP, van der Meche FG, Schmitz PI. Interobserver agreement in the assessment of muscle strength and functional abilities in Guillain-Barre syndrome. Muscle Nerve. 1991 Nov;14(11):1103-9. doi: 10.1002/mus.880141111. PMID 1745285
- [Background] Merkies IS, Kieseier BC. Fatigue, Pain, Anxiety and Depression in Guillain-Barre Syndrome and Chronic Inflammatory Demyelinating Polyradiculoneuropathy. Eur Neurol. 2016;75(3-4):199-206. doi: 10.1159/000445347. Epub 2016 Apr 15. PMID 27077919
- [Background] Borg GA. Psychophysical bases of perceived exertion. Med Sci Sports Exerc. 1982;14(5):377-81. PMID 7154893
- [Background] Andrews AW, Middleton A. Improvement During Inpatient Rehabilitation Among Older Adults With Guillain-Barre Syndrome, Multiple Sclerosis, Parkinson Disease, and Stroke. Am J Phys Med Rehabil. 2018 Dec;97(12):879-884. doi: 10.1097/PHM.0000000000000991. PMID 29952780
- [Background] Mong Y, Teo TW, Ng SS. 5-repetition sit-to-stand test in subjects with chronic stroke: reliability and validity. Arch Phys Med Rehabil. 2010 Mar;91(3):407-13. doi: 10.1016/j.apmr.2009.10.030. PMID 20298832
- [Background] Ferreira PL, Ferreira LN, Pereira LN. [Contribution for the validation of the Portuguese version of EQ-5D]. Acta Med Port. 2013 Nov-Dec;26(6):664-75. Epub 2013 Dec 20. Portuguese. PMID 24388252
- [Background] Langer D, Charususin N, Jacome C, Hoffman M, McConnell A, Decramer M, Gosselink R. Efficacy of a Novel Method for Inspiratory Muscle Training in People With Chronic Obstructive Pulmonary Disease. Phys Ther. 2015 Sep;95(9):1264-73. doi: 10.2522/ptj.20140245. Epub 2015 Apr 9. PMID 25858974
- [Background] Jung JH, Kim NS. The effect of progressive high-intensity inspiratory muscle training and fixed high-intensity inspiratory muscle training on the asymmetry of diaphragm thickness in stroke patients. J Phys Ther Sci. 2015 Oct;27(10):3267-9. doi: 10.1589/jpts.27.3267. Epub 2015 Oct 30. PMID 26644689
- [Background] Angst F, Aeschlimann A, Angst J. The minimal clinically important difference raised the significance of outcome effects above the statistical level, with methodological implications for future studies. J Clin Epidemiol. 2017 Feb;82:128-136. doi: 10.1016/j.jclinepi.2016.11.016. Epub 2016 Dec 14. PMID 27986610